CLINICAL TRIAL: NCT02242578
Title: Effect of rTMS Over the Medial Cerebellum on Negative Symptoms and Cognitive Dysmetria in Subjects With Treatment Refractory Schizophrenia
Brief Title: Treating Refractory Schizophrenia With rTMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB approval expired and study ceased.
Sponsor: Seton Healthcare Family (Other)
Collaborators: Abbott Medical Devices (Industry); University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Robert J. Buchanan, Chief of Functional and Restorative Neurosurgery and Neurosciences, Seton Healthcare Family
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-11-149
Record Dates: First submitted 2014-09-12; First posted 2014-09-17 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Schizophrenia
Keywords: Negative symptoms
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Active rTMS stimulation (1 Hz rTMS, 10 Hz rTMS)
  Interventions: Device: 1 Hz rTMS; Device: 10 Hz rTMS
- Placebo (Experimental): Sham rTMS stimulation (1 Hz rTMS, 10 Hz rTMS)
  Interventions: Device: 1 Hz rTMS; Device: 10 Hz rTMS

INTERVENTIONS:
Device: 1 Hz rTMS — About 1,000 stimulation pulses over 20 min
Device: 10 Hz rTMS — About 1,000 stimulation pulses over 20 min

SUMMARY:
Symptomatic treatment of the negative symptoms in schizophrenia (such as social withdrawal, affective flattening, poor motivation, and apathy) with medications and psychotherapy are almost non-existent, whereas treatment of the positive symptoms (hallucinations and delusions) has been more effective with psychotropic medications. The proposed research on human subjects using a non-invasive technology (such as repetitive transcranial magnetic stimulation [rTMS]) will provide efficacy data for treating negative symptoms.

The hypotheses are that 1) Cerebellar stimulation will cause activation of thalamic and frontal cortical networks associated with attentional processes as a component of the "distracted" affect of schizophrenia; 2) Cerebellar stimulation will cause activation of the reticular activating system (RAS), and this will allow the "mutism", which is a negative symptom, to be partially improved.

DETAILED DESCRIPTION:
Background and Significance

There is increasing evidence from neuropsychological and imaging studies that cerebellar function is relevant not only to motor coordination, but equally to cognition and behavior (Rapoport et al., 2000). Selective modulation of cerebello-thalamocortical pathways, in turn, is believed to provide an additional means of modulating cortical function. Repetitive transcranial magnetic stimulation (rTMS) can modulate cortical excitability focally in conscious subjects. Trains with slow frequency (i.e.,1 Hz) are known to suppress cortical excitability (Chen et al., 1997), whereas facilitation occurs if frequencies higher than 5 Hz are used (Berardelli et al., 1998). With respect to rTMS of the cerebellum, a major impact on cognitive function (Oliveri et al., 2007) has been described.

The cerebellum is a very good candidate to be the generator for intracortical inhibition; its stimulation can modulate the cortical inhibition. Invasive studies by Robert Heath at Tulane University revealed that the cerebellum is strongly connected to 2 structures at the core of the proposed abnormal circuitry in schizophrenia, the septal nuclei and the hippocampus (HC). According to his theory and findings, the septal nuclei are involved in positive mood regulation, pleasure. The firing of the HC was correlated with negative affect and sadness (Heath et al, 1980). By stimulating the fastigial nucleus and vermis of the cerebellum, the septal nuclei were facilitated to fire and the HC was inhibited. The other component of what Heath referred to as the "aversive system", the amygdala was also inhibited. This central role of the cerebellum in this circuit is analogous to its role in "smoothing" the flow of movements. When considering emotion and cognition, the cerebellum has a smoothing function. Aside from direct monosynaptic connections between these sites, there is evidence that the deep cerebellar nuclei are connected to the parietal cortex, temporal cortex, as well as the cingulate gyrus. These are all areas that have limbic function. The cerebellum is also directly connected to the midbrain reticular activating system (RAS). This region is responsible for levels of consciousness and arousal. By potentiating the activation of the RAS, wthe investigators e can increase the decreased level of arousal, which in many schizophrenia patients is akin to psychomotor retardation and mutism (catatonic). Midline deep cerebellar nuclei efferents have been traced to the hypothalamus, central nuclei of the thalamus, which are also associative (cognitive) and limbic in function. The Locus Ceruleus and the substantia nigra, in the brain stem are also monosynaptically connected to the cerebellum.

The cerebellum is connected to thalamus and motor cortex (frontal cortex) through cerebello-thalamo-cortical pathway. And as stated above it is also connected to a vast array of limbic structures, making it a good choice to use to modulate abnormal activity in these structures.

Purkinje cells, the output neurons of cerebellar cortex reduce the excitatory drive from the deep cerebellar nuclei via the ventrolateral thalamus to inhibitory neurons in the motor cortex. Activation of Purkinje cells will inhibit the thalamic drive to intracortical inhibitory neurons, therefore, decrease the intracortical inhibitory interneuron activity and decrease in SICI and CSP. On the other hand, inhibition of Purkinje cerebellar cells is expected to have opposite effect and release the thalamus from inhibitory control, increase the thalamic drive to stimulate the inhibitory interneurons which can be demonstrated by increase in SICI and CSP Indeed, applying inhibitory rTMS at frequency of 1 Hz resulted in increase in SICI (Langguth et al., 2008).

The midline deep cerebellar nuclei, those that are anatomically and phylogenetically related to the vermis, also send collaterals to the reticular activating system (RAS) of the brain stem. By increasing the excitatory (Glu) drive on the RAS, the subject will experience increased awareness and connection to their environment.

For decades, the cerebellum has been thought to be predominantly involved in motor performance and cognitive operations. Recently, however, a growing body of evidence indicates that the cerebellum is also involved in emotion. The first evidence for cerebellar involvement in emotion came from the work of Robert G. Heath during the early fifties. Although his initial work predominantly involved the electrical stimulation of the septum, he then began research on stimulation of the cerebellum, thinking that it might provide a better entry to the emotional circuitry of the brain. Several cerebellar pacemaker studies by Heath did indeed demonstrate positive effects on mood and personality in patients with psychiatric illness after electrical stimulation of the cerebellum. Moreover, Schmahmann and Sherman provided clinical support for the role of the cerebellum and particularly the vermis in the regulation of emotion and mood. Given its modulatory role on emotion, the midline cerebellar vermis together with the fastigial nucleus and the flocculonodular lobe have been designated the limbic cerebellum (Schutter and van Honk 2005). Furthermore, additional evidence for the involvement of the cerebellum in schizophrenia was supported by genetic, structural and functional imaging data (Sandyk et al., 1991; Nopoulos et al., 1999; Ichimiya et al., 2001; Varnas et al., 2007) as well as by clinical evidence (Deshmukh et al., 2002; Ho et al., 2004; Varambally et al., 2006). For example, in an animal model for schizophrenia using prenatal infection of mice with human influenza virus, the animal developed behavioral changes similar to those of schizophrenia and was associated with altered expression of cerebellar genes (Fatemi et al., 2008). Some studies reported smaller bilateral cerebellar volumes as compared to controls in first episode schizophrenia patients (Bottmer et al., 2005). One of the first studies to demonstrate the importance of a dysfunctional cerebellar circuitry in schizophrenia was a positron emission tomography (PET) study (Andreasen et al., 1996). The authors examined memory performance in schizophrenia patients and correlate it to blood flow in cerebello-thalamo-cortical pathway. They used two tasks for memory, namely an easy and a relatively difficult one. While patients with schizophrenia showed normal performance on the easy practiced memory task they already demonstrated decreased blood flow in the cerebello-thalamo-cortical pathway. By contrast, in the relatively more difficult memory task, schizophrenia patients performed worse than healthy controls and displayed significantly lowered frontal and cerebellar blood flow (Andreasen et al., 1996).

Consistent with the assumed disruption of the cerebellothalamo- cortical pathway in schizophrenia is evidence from two proton magnetic resonance spectroscopic imaging (HMRS) studies. Lower levels of N-acetylaspartate (NAA), a marker for neuron density and viability, were found in the thalamus and cerebellar vermis (Deicken et al., 2001) in patients with schizophrenia. In keeping with these findings, lower NAA levels in the vermis and cerebellar cortex have also been found (Ende et al., 2005) as well as in mediodorsal region of the thalamus (Ende et al., 2001). In addition, poor executive functioning in patients with schizophrenia was associated with volumetric reductions in the cerebello-thalamo-cortical network (Rusch et al., 2007). Moreover, a diffusion tensor imaging (DTI) study has shown that patients with schizophrenia demonstrate abnormality in the connectivity between cerebellum and thalamus with possible difference between the right and left cerebellum (Magnota et al., 2008). Investigating connectivity between the cerebellum and thalamus in schizophrenia using diffusion tensor tractography: A pilot study). Another DTI study found neuronal disorganization in the superior peduncle with neuronal disorganization being associated with poor cognitive performance (Okugawa et al., 2006). Finally, the activity of right and left cerebellum may not be the same. For example, impaired working memory in schizophrenia is associated with over and under-activation along the cerebellothalamo- cortical pathway with under-activation of the left DLPFC and right cerebellum and over-activation of the left cerebellum (Mendrek et al., 2005).

To date, cerebellar involvement in schizophrenia remains a subject of ongoing study. It was shown that motor impairments in schizophrenia are related to cerebellar malfunction. Several studies report that the cerebellum is indeed involved in cognitive (Eyler et al., 2004; Aasen et al., 2005; Kiehl et al., 2005) and affective (Paradiso et al., 2003; Takahashi et al., 2004; Stip et al., 2005) impairments. This study aims to clarify the role of the cerebellum in development of negative symptoms through its regulation of cortical inhibition, activation of the septal region with reciprocal inactivation of the hippocampus, and RAS activation.

Experimental Design and Methods/Procedures

1. rTMS over the vermis of the cerebellum
2. 5 sessions/week for 1 week
3. Randomization as explained below.

Patients will be randomly assigned to either the high frequency or low frequency Medial Cerebellum Target Treatment protocol. Each group will then be entered into a randomized, double-blind, sham-controlled, parallel-design clinical trial that consists of three main phases: (1) Baseline Psychiatric and Psychometric Testing Exam; (2) 5 rTMS treatments, double-blind, in 5 treatment sessions/week with active or sham rTMS for over a period of 1 week; and (3) a follow-up period of 3 weeks. The patients will then be reassigned to the other Frequency (either high or low) Arm of the study. The protocol will then be repeated. Patients and the investigators, except the investigator who applied rTMS, will be blinded to the treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolling to the study:

  * must be stable on their medications at the start of their enrollment in the study and throughout the duration of the study;
  * must have no history of substance use of substance-dependence issues over at least the past six months;
  * must be able to and have the capacity to provide consent;
  * and if older patient, he/she must be able to participate without a safeguard to be present.

Exclusion Criteria:

* Patients excluded from the study are:

  * Patients with typical clinical considerations that exclude them from treatment with TMS (i.e., patients who have had head injuries, patients with metal implants, patients with a history of seizures, patients with elevated risk of seizures, patients who are taking medications that may interfere with TMS or potentiate the related side effects, etc.).
  * Patients who have had changes in their medications (i.e., patients must be stable on their medications throughout their participation in the study).
  * Patients with history of substance abuse or substance-dependence anytime over the past six months.
  * Patients who are unable (i.e., do not have the capacity) to consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01-24 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Buchanan, MD, Principal Investigator — Seton Family Hopsitals
Locations (1):
- Seton Brain and Spine Institute "Brain Stimulation Laboratory", Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreasen NC, O'Leary DS, Cizadlo T, Arndt S, Rezai K, Ponto LL, Watkins GL, Hichwa RD. Schizophrenia and cognitive dysmetria: a positron-emission tomography study of dysfunctional prefrontal-thalamic-cerebellar circuitry. Proc Natl Acad Sci U S A. 1996 Sep 3;93(18):9985-90. doi: 10.1073/pnas.93.18.9985. PMID 8790444
- [Background] Ende G, Hubrich P, Walter S, Weber-Fahr W, Kammerer N, Braus DF, Henn FA. Further evidence for altered cerebellar neuronal integrity in schizophrenia. Am J Psychiatry. 2005 Apr;162(4):790-2. doi: 10.1176/appi.ajp.162.4.790. PMID 15800155
- [Background] Ho BC, Mola C, Andreasen NC. Cerebellar dysfunction in neuroleptic naive schizophrenia patients: clinical, cognitive, and neuroanatomic correlates of cerebellar neurologic signs. Biol Psychiatry. 2004 Jun 15;55(12):1146-53. doi: 10.1016/j.biopsych.2004.02.020. PMID 15184033
- [Background] Nopoulos PC, Ceilley JW, Gailis EA, Andreasen NC. An MRI study of cerebellar vermis morphology in patients with schizophrenia: evidence in support of the cognitive dysmetria concept. Biol Psychiatry. 1999 Sep 1;46(5):703-11. doi: 10.1016/s0006-3223(99)00093-1. PMID 10472423
- [Background] Picard H, Amado I, Mouchet-Mages S, Olie JP, Krebs MO. The role of the cerebellum in schizophrenia: an update of clinical, cognitive, and functional evidences. Schizophr Bull. 2008 Jan;34(1):155-72. doi: 10.1093/schbul/sbm049. Epub 2007 Jun 11. PMID 17562694
- [Background] Rusch N, Spoletini I, Wilke M, Bria P, Di Paola M, Di Iulio F, Martinotti G, Caltagirone C, Spalletta G. Prefrontal-thalamic-cerebellar gray matter networks and executive functioning in schizophrenia. Schizophr Res. 2007 Jul;93(1-3):79-89. doi: 10.1016/j.schres.2007.01.029. Epub 2007 Mar 26. PMID 17383859
- [Background] Rapoport M, van Reekum R, Mayberg H. The role of the cerebellum in cognition and behavior: a selective review. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):193-8. doi: 10.1176/jnp.12.2.193. PMID 11001597

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated and no data collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Scores at 1 Week
Description: Participants will receive baseline and post-treatment protocol neuropsychiatric measures. These rating scales are accepted and standardized.
Time Frame: Participants will be followed for an expected average of 5 weeks
Population: Study was terminated (that is, stopped prematurely) and no data were collected for one or more Outcome Measures.
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in Electroencephalographic (EEG) Measures at 1 Week
Description: Electroencephalographic (EEG) recordings and evaluations:
  Patients will undergo 19-channel EEG recordings before, and immediately after the end of the 5-day rTMS treatment. Patients will be kept awake during this procedure to control for the effects of sleep on EEG. Each EEG recording will be performed by employing scalp electrodes placed according to the International 10-20 system. Data will be analyzed for changes in the spectral characteristics of the EEG, most importantly in delta and beta frequency bands.
Time Frame: Participants will be followed for an expected average of 5 weeks
Population: Study was terminated (that is, stopped prematurely) and no data were collected for one or more Outcome Measures.
Arm/Group | Active | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 0 year
Description: Study terminated, no data collected.
Arm/Group | Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study was terminated and no data was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT02242578/Prot_SAP_000.pdf